CLINICAL TRIAL: NCT02727387
Title: Study With High Doses of Chemotherapy, Radiotherapy and Consolidation Therapy With Ciclofosfamide and Anticyclooxygenase 2, for the Metastatic Ewing Sarcoma
Brief Title: Protocol for the Treatment of Metastatic Ewing Sarcoma
Acronym: EW-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG/AIEOP EW-2
Record Dates: First submitted 2016-03-23; First posted 2016-04-04 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Ewing's Sarcoma (ES)
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Temozolomide; Irinotecan; Doxorubicin; Ifosfamide; Cyclophosphamide; Etoposide; Busulfan; Melphalan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEMIRI+VIN+ADM+IFO+ CYC+ETO+BUMEL (Experimental): 2cycles of Temozolomide(500 mg/m2)+Irinotecan(250 mg/m2) and 2cycles of Vincristine(1.4mg/m2)+ Adriamycin(90mg/m2)+Ifosfamide (9gr/m2) alternes with 2 cycles of Ciclofosfamide(4g/m2)+Etoposide (600mg/m2) followed by radiotherapy (42-54 Gy) and 2cycles of Ifosfamide (9gr/m2) + Etoposide(300mg/m2) alternes with to 2cycles of Vincristine (1.4mg/m2)+ Adriamycin (80mg/m2)+ Ciclofosfamide(1.2g/m2) and Busulfan(0.8-1.2 mg/Kg)+Melfalan(140 mg/m2)+PBSCT and 6 months with Celecoxib (500mg/m2/die for<14 years old ,800 mg/die for>14 years old) Ciclofosfamide (oral therapy 35mg/m2/die for<14 years old, 50 mg/m2 for>14 years old)
  Interventions: Drug: TEMIRI; Drug: ADM; Drug: IFO; Drug: CYC; Drug: ETO; Drug: BUMEL; Drug: VIN

INTERVENTIONS:
Drug: TEMIRI — Window therapy frontline for VHR patients
  Other Names: Temozolomide + Irinotecan
Drug: ADM — Drug used in the Induction phase in association with Vincristine, Ifosfamide, cyclophosphamide and Etoposide
  Other Names: Adriamycin
Drug: IFO — Drug used in the Induction phase in association with Vincristine, Adriamycin, cyclophosphamide and Etoposide
  Other Names: Ifosfamide
Drug: CYC — Drug used in the Induction phase in association with Vincristine, Ifosfamide, Adriamycin and Etoposide
  Other Names: Cyclophosphamide
Drug: ETO — Drug used in the Induction phase in association with Vincristine, Ifosfamide, cyclophosphamide and Adriamycin
  Other Names: Etoposide
Drug: BUMEL — Consolidation phase
  Other Names: busulfan + melphalan
Drug: VIN — Drug used in the Induction phase in association with cyclophosphamide , Ifosfamide, Adriamycin and Etoposide
  Other Names: Vincristine

SUMMARY:
Study for the treatment of metastatic Ewing sarcoma with high doses chemotherapy, radiotherapy and maintenance therapy.

DETAILED DESCRIPTION:
Study for the treatment of Ewing metastatic sarcoma with and induction phase with Vincristine (VIN), Adriamycin (ADM), Ciclofosfamide(CYC), Ifosfamide(IFO), Etoposide(ETO) and radiotherapy (RT)followed by a consolidation phase with Busulfan and Melfalan (BUMEL) and Peripheral Blood Stem Cells Transplantation (PBSCT) and a subsequent maintenance phase with Ciclofosfamide and Celecoxib for High Risk (HR) patients.

Very High Risk (VHR) patients will receive a prior frontline therapy with Temozolomide and Irinotecan (TEMIRI), while patient with lung metastasis only will undergo to total lung irradiation after PBSCT

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Ewing's sarcoma
* Age ≤ 40 years
* No previous treatment
* Multiple skeletal metastasis or bone marrow infiltration , with/without lung/pleural metastasis
* Signed Informed Consent

Exclusion Criteria:

* Localized Ewing's sarcoma
* Any contraindications to the study treatment
* Female patients who not accept to use an effective birth control method.
* Pregnant or breast-feeding patients

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Expected average 3 year
  Evaluation of the OS in patients treated according to the protocol
Event Free Survival (DFS) | Expected average 1 year
  Evaluation of the time in which the patient do not experience any progression, relapse of toxicity event when treated according to the protocol

SECONDARY OUTCOMES:
Safety - Incidence and grade of treatment-emergent Adverse Events | every 21 days up to 1 year
  Incidence and grade of treatment-emergent Adverse Events
Evaluation of Quality of life using Pediatric Quality of Life Inventory (PedQL) -in child and adolescents(EORTC QLQ-C30) for children and adolescents | every 3 weeks for the first 6 months and 3 monthly up to 1 year
  Evaluation of patient's Quality of life: comparison of the Baseline and On treatrment quality of life score using PedQL
Evaluation of Quality of life using European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients (EORTC QLQ-C30) for adult patients | every 3 weeks for the first 6 months and 3 monthly up to 1 year
  Evaluation of patient's Quality of life: comparison of the Baseline and On treatrment quality of life score using EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Luksch, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (13):
- Italy (13):
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Azienda ospedaliero universitaria consorziale policlinico - bari, Bari
  - Istituto Ortopedico Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna
  - Servizio di Oncoematologi Pediatrica Ospedale microcitemico ASL 8, Cagliari
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS INT Milano, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Ospedale Pediatrico Bambin Gesu', Roma
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Picci P, Bohling T, Bacci G, Ferrari S, Sangiorgi L, Mercuri M, Ruggieri P, Manfrini M, Ferraro A, Casadei R, Benassi MS, Mancini AF, Rosito P, Cazzola A, Barbieri E, Tienghi A, Brach del Prever A, Comandone A, Bacchini P, Bertoni F. Chemotherapy-induced tumor necrosis as a prognostic factor in localized Ewing's sarcoma of the extremities. J Clin Oncol. 1997 Apr;15(4):1553-9. doi: 10.1200/JCO.1997.15.4.1553. PMID 9193352
- [Background] Gardner SL, Carreras J, Boudreau C, Camitta BM, Adams RH, Chen AR, Davies SM, Edwards JR, Grovas AC, Hale GA, Lazarus HM, Arora M, Stiff PJ, Eapen M. Myeloablative therapy with autologous stem cell rescue for patients with Ewing sarcoma. Bone Marrow Transplant. 2008 May;41(10):867-72. doi: 10.1038/bmt.2008.2. Epub 2008 Feb 4. PMID 18246113
- [Background] Paulussen M, Ahrens S, Burdach S, Craft A, Dockhorn-Dworniczak B, Dunst J, Frohlich B, Winkelmann W, Zoubek A, Jurgens H. Primary metastatic (stage IV) Ewing tumor: survival analysis of 171 patients from the EICESS studies. European Intergroup Cooperative Ewing Sarcoma Studies. Ann Oncol. 1998 Mar;9(3):275-81. doi: 10.1023/a:1008208511815. PMID 9602261